CLINICAL TRIAL: NCT02037100
Title: Sleep Disordered Breathing and Impaired Glucose Homeostasis in Obese Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Schneider Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TASMC-14-RT-07-066-CTIL
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: SDB; T2DM; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- T2DM: Children 6-20 years old diagnosed with T2DM
- Obesity

SUMMARY:
SDB has been identified as an important risk factor for insulin resistance and the metabolic syndrome.

In a recent study in patients with SDB and T2DM it was shown that CPAP therapy can lead to improvements in postprandial glucose levels and in glycosylated hemoglobin levels (HbA1c).

In children, there are only 3 studies that have examined the relations between SDB, obesity and the metabolic syndrome.

In order to further understand the relative contribution of SDB to the development of impaired glucose homeostasis and metabolic abnormalities we aim to investigate the prevalence and severity of SDB in children with T2DM compared to obese children without T2DM. The investigators hypothesize that SDB will be more prevalent and more severe among obese children with T2DM compared with the general obese pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with T2DM
* obese

Exclusion Criteria:

-

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children 6-20 years old
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-06; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Investigate the prevalence and severity of SDB among children with T2DM compared to its prevalence in non-diabetic obese children. | In 6 months
To measure markers of inflammation and oxidative stress known to be associated with cardiovascular morbidity in children with T2DM and SDB compared to non-diabetic obese children. | In 6 months
To examine changes in metabolic measures and markers of inflammation and oxidative stress in response to treatment for SDB (adenotonsillectomy) in children with T2DM compared to obese children without T2DM. | In 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel